CLINICAL TRIAL: NCT01716962
Title: Effects of Positive End-expiratory Pressure and Tidal Volume on Fluid Responsiveness of Acute Respiratory Distress Syndrome.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Huang chung chi, Director of Department of Respiratory Therapy, Chang Gung University, Chang Gung Memorial Hospital
Other Study IDs: CGMF IRB 100-4473A3
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute respiratory distress syndrome, Fluid responsiveness, Pulse pressure variation; Pleth variability index, Passive leg raising test
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARDS with acute circulatory failure: acute respiratory distress syndrome with acute circulatory failure with infusion of 6% tetrastarch for a total of 500ml
  Interventions: Other: Infusion of 6% tetrastarch for a total of 500 ml

INTERVENTIONS:
Other: Infusion of 6% tetrastarch for a total of 500 ml

SUMMARY:
Fluid responsiveness (FR)refers to the ability of heart to increase its stroke volume in response to volume load.Low tidal volume and high PEEP exerts contrast effect on the prediction of fluid responsiveness, the aim of this study is to compare the relative predicting power of the dynamic preload indicator (PPV, SVV), passive leg raising test, and pleth variability index (PVI) on the fluid responsiveness of acute respiratory distress syndrome ventilated with various PEEP levels or various tidal volumes.

DETAILED DESCRIPTION:
In septic critically ill mechanically ventilated patients with acute circulatory failure, inadequate volume resuscitation leads to multiple organ failure. Early goal-directed therapy emphasizes early and aggressive hemodynamic support in patients with severe sepsis and septic shock. On the other hand, because of increased microvascular permeability and capillary leakage, conservative fluid management and more aggressive restriction in fluid accumulation to reduce lung water and tissue edema has been suggested by acute respiratory distress syndrome net. Fluid responsiveness refers to the ability of the heart to increase its stroke volume in response to volume load. Accurately predicting volume responsiveness will be beneficial in obviating the need for unnecessary fluid loading, and in detecting patients who may benefit from a volume load.

By inducing cyclic changes in pleural and transpulmonary pressure, mechanical ventilation results in cyclic changes in the preload and afterload, and therefore, the cyclic variation in systolic and pulse pressure. Recently, a systemic review concluded that dynamic preload indicator [pulse pressure variation (PPV), stroke volume variation (SVV)] are highly accurate in predicting volume responsiveness in critically ill patients. However, this technique is limited to patients who receive controlled ventilation with adequate tidal volume (> 8 ml/Kg) and sedation or paralysis is needed to abolish the spontaneous ventilation.

For acute respiratory distress syndrome patients, protective ventilatory strategy suggested low tidal volume to 6 ml/Kg. On the contrary, high PEEP needed for acute respiratory distress syndrome to prevent VALI induces a leftward shift to the steep pat of the Frank-Starling curve and increase the fluid responsiveness. Whether the dynamic preload indicators (PPV and SVV) are still effective in acute respiratory distress syndrome patients for predicting fluid responsiveness remain controversial.

Passive leg raising (PLR), by inducing a gravitational transfer of blood from the lower part of the body toward the central circulatory compartment, can be considered as a brief "self volume challenge". Recently, a systemic review and meta-analysis concluded that PLR-induced changes in cardiac output reliably predict fluid responsiveness regardless of ventilation mode, underlying cardiac rhythm and technique of measurement and can be recommended for routine assessment of fluid responsiveness in the majority of ICU population. More importantly, this prediction remains very valuable in patients with cardiac arrhythmias or spontaneous breathing activity.

Respiratory variations in the pulse oximeter plethysmographic waveform amplitude (ΔPOP) have been shown to be able to predict fluid responsiveness in mechanically ventilated patients. The main advantage of this index is that it is noninvasive, widely available, and inexpensive. Perfusion index (PI), the percentage between the infrared pulsatile and nonpulsatile signal, reflects the amplitude of the pulse oximeter waveform. Recently, Pleth Variability Index (PVI), derived from perfusion index, affords a continuous monitoring of ΔPOP. PVI has been shown to be correlated to ΔPOP and PPV and has been demonstrated to be equivalent to SVV as a predictor of fluid responsiveness in ventilated patients during major surgery. However, whether the PVI can predict the fluid responsiveness in acute respiratory distress syndrome necessitating low tidal volume and high PEEP is not clear.

Because of the aforementioned contrasting effects of low tidal volume and high PEEP on the prediction of fluid responsiveness, the aim of this study is to compare the relative predicting power of the dynamic preload indicator (PPV, SVV), passive leg raising test, and PVI on the fluid responsiveness of acute respiratory distress syndrome ventilated with various PEEP levels or various tidal volumes.

ELIGIBILITY:
Inclusion Criteria: Clinical signs of inadequate tissue perfusion were defined

1. systolic blood pressure< 9 mmHg(or a decrease > 50 mmHg in previously hypertensive patients)
2. need of vasopressive drugs(dopamine > 5 ug/Kg/min or norepinephrine)
3. urine output<0.5 mL/Kg/hr for at least 2 hrs
4. tachycardia (heart rate >100/min)
5. presence of skin mottling.

Exclusion Criteria:

1. patient with spontaneous respiratory activity
2. cardiac arrhythmia
3. known intracardiac shunt
4. contraindication for passive leg raising(PLR),e.g.,pelvic trauma
5. unstable spine injuries or leg amputation
6. hemodynamic instability during the procedure,defined by a variation in heart rate or blood pressure of>10%over the 15-min period before starting the protocol
7. Patients of renal failure necessitate renal replacement therapy will be excluded also.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated ALL/ARDS patients conforming to the American European Consensus Conference criteria with acute circulatory failure for whom the attending clinician had decided to administer fluid will be enrolled.This decision was based on the presence of at least one clinical sign of inadequate tissue perfusion in the absence of contraindication for fluid infusion.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
increase of cardiac output after volume expansion | 4 hours
  Patients are classified to be volume expansion responders or nonresponders according to whether the volume expansion induced cardiac index increase at the end of hydroxyethyl starch infusion is ≧15% or < 15% of baseline cardiac index.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Chi Huang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan, Taiwan